CLINICAL TRIAL: NCT00099944
Title: Efficacy and Safety of Vildagliptin in Combination With Glimepiride in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLAF237A2305
Record Dates: First submitted 2004-12-21; First posted 2004-12-22 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- LAF237 50 mg qd + glimepiride 4 mg qd (Experimental): LAF237 50 mg qd + glimepiride 4 mg qd
  Interventions: Drug: vildagliptin; Drug: Glimepiride
- LAF237 50 mg bid + glimepiride 4 mg qd (Experimental): LAF237 50 mg bid + glimepiride 4 mg qd
  Interventions: Drug: vildagliptin; Drug: Glimepiride
- LAF237 placebo + glimepiride 4 mg qd (Placebo Comparator): LAF237 placebo + glimepiride 4 mg qd
  Interventions: Drug: Glimepiride; Drug: LAF237 placebo

INTERVENTIONS:
Drug: vildagliptin
  Arms: LAF237 50 mg bid + glimepiride 4 mg qd; LAF237 50 mg qd + glimepiride 4 mg qd
Drug: Glimepiride — Glimepiride 4 mg qd
Drug: LAF237 placebo
  Arms: LAF237 placebo + glimepiride 4 mg qd

SUMMARY:
Many people with type 2 diabetes cannot maintain target blood glucose levels when taking a single oral drug. The purpose of this study is to assess the safety and effectiveness of two doses of vildagliptin, an unapproved drug, in lowering overall blood glucose levels when added to glimepiride in people with type 2 diabetes not at target blood glucose levels on a sulfonylurea alone.

ELIGIBILITY:
Inclusion Criteria:

* Blood glucose criteria must be met
* Previously treated with a sulfonylurea for at least 3 months
* Body mass index (BMI) in the range 22-45

Exclusion Criteria:

* Type 1 diabetes
* Pregnancy or lactation
* Evidence of serious cardiovascular complications
* Evidence of serious diabetic complications
* Laboratory value abnormalities as defined by the protocol
* Known sensitivity to glimepiride
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2004-05; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c after 24 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose at 24 weeks
Patients with endpoint HbA1c <7% after 24 weeks
Patients with reduction in HbA1c >/=to 0.7% after 24 weeks
Adverse event profile after 24 weeks of treatment
Change from baseline in HbA1c at 24 weeks for patients with high baseline HbA1c vs. low baseline HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Garber AJ, Foley JE, Banerji MA, Ebeling P, Gudbjornsdottir S, Camisasca RP, Couturier A, Baron MA. Effects of vildagliptin on glucose control in patients with type 2 diabetes inadequately controlled with a sulphonylurea. Diabetes Obes Metab. 2008 Nov;10(11):1047-56. doi: 10.1111/j.1463-1326.2008.00859.x. Epub 2008 Feb 18. PMID 18284434